CLINICAL TRIAL: NCT01401504
Title: A Phase I, Non-randomized, Open-label, Repeat Oral Administration Study of ASP3026 in Patients With Solid Tumors
Brief Title: Study of an Investigational Drug, ASP3026, in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3026-CL-0102
Record Dates: First submitted 2011-06-30; First posted 2011-07-25 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Solid Tumor
Keywords: Anti-cancer; ASP3026; Anaplastic Lymphoma Kinase (ALK)
MeSH Terms: interventions — ASP3026

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASP3026 (Experimental)
  Interventions: Drug: ASP3026

INTERVENTIONS:
Drug: ASP3026 — oral

SUMMARY:
A study to evaluate the safety and anti-tumor activity of ASP3026 in patients with advanced malignancies (solid tumors).

DETAILED DESCRIPTION:
This study will be conducted using a traditional 3 + 3 dose escalation study design. Enrollment of at least 3 subjects is planned for each dosing cohort. The decision to expand a cohort or dose escalate will be based on the occurrence of dose limiting toxicities (DLTs) in Cycle 1 that are considered by the Investigator to be related (possibly or probably) to ASP3026. The Safety Data Review Committee may elect to enroll additional subjects in a cohort to further evaluate the dose level. Each cycle will include 28 days of continuous dosing with ASP3026. Treatment with ASP3026 may continue until one of the discontinuation criteria is met.

The maximum tolerated dose (MTD) is defined as the highest dose of ASP3026 on a dosing schedule at which < 33% of subjects experience a DLT during Cycle 1. The MTD or lower dose, as determined by the Safety Data Review Committee, will be the recommended Phase 2 dose (RP2D). Twelve additional patients will be treated at the RP2D to further evaluate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Histologically or cytologically confirmed diagnosis of a relapsed/refractory solid tumor
* Patient meets at least 1 of the following criteria:

  * Disease progression despite standard therapies
  * No standard therapies are available or such therapies are not anticipated to result in a durable response
  * Standard therapies are considered unsuitable or have been refused
* Life expectancy > 12 weeks
* Able to be hospitalized from 1 day prior to the initial dosing until day 15 of the dosing, and from day 27 until day 29 of the dosing

Exclusion Criteria:

* Patient exhibits persistent subjective and objective findings of toxicity ≥ Grade 2 (CTCAE v4.0-JCOG) from the previous cancer treatment with antitumor effect (except of alopecias)
* Received previous treatment with antitumor effect within 21 days prior to the scheduled initial dosing
* Patient had a major surgical procedure within 21 days prior to the scheduled initial dosing or a major surgical procedure scheduled during the course of the study
* Use of an investigational drug or device within 21 days prior to the scheduled initial dosing
* Use of blood transfusion or hematopoietic growth factors within 14 days prior to the scheduled initial dosing
* A positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV)
* Known history of a positive test for human immunodeficiency virus (HIV) infection
* Patient has central nervous system (CNS) or leptomeningeal involvement with clinical symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ASP3026 assessed by recording of adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) and clinical observations | Up to 30 days after last subject discontinues treatment

SECONDARY OUTCOMES:
Pharmacokinetics of ASP3026 by assessment of area under the curve over the time (AUC) and maximum concentration (Cmax) in plasma and urine | Up to Day 29
Objective response rate (ORR) | 30 Days after the last subject discontinues treatment
  Objective response rate is the proportion of subjects who experience complete response/remission (CR) or partial response/remission (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kansai, Japan

REFERENCES:
- [Derived] Ono A, Murakami H, Seto T, Shimizu T, Watanabe S, Takeshita S, Takeda K, Toyoshima J, Nagase I, Bahceci E, Morishita M, Morita S, Fukuoka M, Nakagawa K. Safety and Antitumor Activity of Repeated ASP3026 Administration in Japanese Patients with Solid Tumors: A Phase I Study. Drugs R D. 2021 Mar;21(1):65-78. doi: 10.1007/s40268-020-00331-2. Epub 2020 Dec 17. PMID 33331996
- [Derived] Ono A, Murakami H, Serizawa M, Wakuda K, Kenmotsu H, Naito T, Taira T, Koh Y, Ohde Y, Nakajima T, Endo M, Takahashi T. Drastic initial response and subsequent response to two ALK inhibitors in a patient with a highly aggressive ALK-rearranged inflammatory myofibroblastic tumor arising in the pleural cavity. Lung Cancer. 2016 Sep;99:151-4. doi: 10.1016/j.lungcan.2016.07.002. Epub 2016 Jul 5. PMID 27565932